CLINICAL TRIAL: NCT04968093
Title: Effect and Feasibility of a Mindfulness-based Treatment for Adolescents Aged 12-18 With Chronic Migraine and High Frequency Episodic Migraine Without Aura
Brief Title: Mindfulness for Adolescents for CM and HFEM
Acronym: MINDKIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MINDKIDS
Record Dates: First submitted 2021-07-13; First posted 2021-07-20 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Migraine in Children; Migraine With Aura
Keywords: Chronic Migraine;; High Frequency Episodic Migraine without Aura;; Mindfulness;; Adolescents
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Intervention Model Description: To assess the impact of a mindfulness-based group treatment for adolescents with CM and HFEM on headache frequency reduction over 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group sessions of mindfulness-based therapy (Other): Education of patients followed by seven group sessions of mindfulness-based therapy
  Interventions: Behavioral: Mindfulness-based therapy.

INTERVENTIONS:
Behavioral: Mindfulness-based therapy. — Educational. Patients are given recommendations on the approach to the use of drugs for acute treatment of migraine headache and on lifestyle issues. Patients will be encouraged to restrict use of acute medications to headaches and to engage in regular physical activity, avoiding skipping meals, remain well hydrated, maintain a regular sleep.
  Mindfulness therapy. The intervention is delivered in small groups and consisted of 7 weekly group sessions. It was aimed to teach and make direct practice with skills intended to enhance sustained, non-judgmental present moment awareness. Each session was conducted by a neurologist and a psychologist. To patients were asked to close their eyes and focus their attention on the breathing so that they can concentrate on the present moment and on all the sensations. Intervention's main topics: posture education; breath use and control; guided body scan; work with sounds; tension release; guided imagery; decentralization of thoughts.

SUMMARY:
Chronic Migraine (CM) and High Frequency Episodic Migraine (HFEM) without Aura affect adolescents' lives in terms of reduced health, reduced ability to perform daily chores and reduced quality of life. The use of pharmacological prophylaxis in these patients warrants caution, whereas the use of behavioral treatments is gaining support in literature.

The main aim of MINDKIDS trial is to test the effect of a seven weekly group sessions of guided mindfulness-based meditation program on 12-month headache frequency reduction, medications intake, disability, anxiety, depression, catastrophizing, and caregivers' burden.

This is a single-arm study. All patients will participate to seven weekly guided sessions (60 minutes each) of guided mindfulness meditation, which is aimed to teach and make direct practice with skills intended to enhance sustained, non-judgmental present moment awareness. The intervention's main topics are: posture education; breath use and control; guided body scan; work with sounds; tension release; guided imagery; decentralization of thoughts. Each session is conducted by a neurologist and a psychologist expert in mindfulness practice. During the sessions, patients are asked to close their eyes and focus their attention on the breathing so that they can concentrate on the present moment and on all the sensations.

Patients were educated to promote a healthy lifestyle: regular physical activity, avoiding skipping meals, hydration, maintain a regular sleep/wake pattern at least 7-8 hours per night.

DETAILED DESCRIPTION:
Background and significance Adolescents with Chronic Migraine (CM) and High Frequency Episodic Migraine (HFEM) without Aura, characterized by 15+ and 9-14 days with headache respectively, pose a relevant burden on adolescents' health, quality of life, as well as on their ability to perform school and leisure time activity. In addition to this, tackling such health conditions in adolescence might be of great importance to reduce the likelihood of a transition to adulthood with CM and medication overuse headache.

In this category of patients, it is suggested to avoid prescribing pharmacological prophylaxis, in favour of non-pharmacological approaches, such as nutraceuticals or behavioural techniques.

Behavioural approaches are considered helpful for younger patients with HFEM and CM to manage pain and to reduce the number of analgesics and the use preventive medications. Mindfulness, in particular, has been applied in several clinical experiences in adults with pain and migraine with encouraging results, with long term benefit similar to that obtained from pharmacological prophylaxis. The clinical use of mindfulness in adolescents is limited to few experiences, however some results in this group of patients are encouraging. A non-randomized pilot study demonstrated acceptability and feasibility of a mindfulness-based treatment for adolescents with recurrent headaches (1). Another study demonstrated how mindfulness was able to reduce depression in children and adolescents suffering from migraine associated with depression (2). A third small pilot study (3) showed positive results with the use of mindfulness in young patients with headache.

Taken as a whole, these studies seem to point out that mindfulness-based protocol for adolescents with CM or HFEM are feasible and acceptable. What has to be better addressed is the effect of such a kind of treatment: available information, however, enable us to hypothesize that reduction in headache frequency from baseline over a 12-months period could be higher or equal to 50%.

ELIGIBILITY:
Inclusion criteria: one of the two main diagnoses are to me met.

1. diagnosis of episodic migraine without aura (code 1.1 of International Classification of Headache Disorders, third version - ICHD-3) at high frequency (HFEM).

   The clinical features are those of code 1.1 of the ICHD-3, with headache lasting 2-72 hours (which is specific to populations aged <18) and with frequency 8-14 days/month for >3 months.
2. Diagnosis of Chronic Migraine (CM) (code 1.3 of International Classification of Headache Disorders, third version). Core features are the following:

   * Headache (migraine-like or tension-type-like1) on 15 days/month for >3 months
   * Headache occurring in a patient who has had at least five attacks fulfilling criteria for Migraine without aura OR for Migraine with aura
   * Headache with migraine-like features for at least 8 days/month for >3 months, i.e. with typical features of migraine with or without aura, or with the headache believed by the patient to be migraine at onset and relieved by a triptan or ergot derivative

Exclusion Criteria:

1. major psychiatric disorders based on clinical history;
2. psychotherapy of any approach in the previous 18 months;
3. previous experience of mindfulness or meditation approach

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Change in headaches frequency as assessed by specific headache diaries in which patient report headaches' presence in each day | 6 and 12 months

SECONDARY OUTCOMES:
Proportion of patients achieving the reduction of 50% or more of days with headache compared to baseline. | 12 months
Change in the number of medications for acute headaches treatment, included in specific headache diaries in which patients indicate the amount of medications consumed to treat headaches | 6 and 12 months
Change in disability scores, assessed with the Pediatric Migraine Disability Assessment (PedMIDAS). | 6 and 12 months
  The PedMIDAS is composed of six items addressing the missed and partially missed school-days, missed and partially missed days for homework activities, missed and partially missed days for leisure activities. The total PedMIDAS score is determined by the sum of items' scores and four severity categories are established: 0-10 no or minimal disability; 11-30 light disability; 31-50 moderate disability; more than 50 high disability
Change in anxiety score, assessed with the Spielberger State-Trait Anxiety Inventory for Children (STAI-CH). | 6 and 12 months
  The STAI-CH is composed by 20 items, rated on a 1-4 scale, which evaluate state anxiety (i.e. temporary feelings at the time of a perceived threat; 0=not at all - 4=very much) and 20 items evaluating trait anxiety (i.e. feelings of stress and worry experienced on a day to day basis; 0=almost never - 4=almost always). The score range is between 20 and 80: higher scores correspond to higher anxiety levels.
Change in depression score, assessed with the Kovacs's Children's Depression Inventory (CDI). | 6 and 12 months
  The CDI consists of 27 items evaluating different symptoms of depression, including mood disturbances, vegetative functions, social behaviour, ability to feel good sensations, self-esteem. The items investigate the influence of depressions in specific contests for young patients. Each item is scored on a 0-2 scale (0=no problem; 1= moderate problem; 2=serious problem) and the total score range is 0-54. A total score higher than 19 indicates risk of depression.
Change in catastrophizing scores, assessed with the Pain Catastrophizing Scale (PCS). | 6 and 12 months
  The PCS addresses the concept of catastrophizing as it relates to pain, i.e. an exaggerated negative mental set brought to bear during actual or anticipated painful experience. It is composed by three subscales each identifying specific dimensions: rumination, which refers to the constant thinking about pain; magnification, which refers to the exaggeration of pain and of its consequences; helplessness, which refers to the belief that there is no or limited possibility that pain may improve. This measure is composed of 13 items, each rated from 0 = "not at all" to 4 = "all the time," yielding total scores ranging from 0 to 52, with higher scores indicating higher tendencies to catastrophize and score values ≥ 30 indicating clinically significant levels of catastrophizing
Change in caregiver burden score, assessed with the Caregiver Burden Inventory (CBI). | 6 and 12 months
  The CBI consists of 24 items evaluated on a 0-4 scale (0=not at all - 4=very much) that describe emotional reactions and difficulties related to the caregiving activity. The items assess issues related to the time required for assistance, the perception of being cut off from other activities and possibilities, fatigue, the reduction of social activities and feelings towards the relative. The total score is linearly transformed on a 0-100 scale: higher scores indicate greater burden.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroalgology Unit, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hesse T, Holmes LG, Kennedy-Overfelt V, Kerr LM, Giles LL. Mindfulness-Based Intervention for Adolescents with Recurrent Headaches: A Pilot Feasibility Study. Evid Based Complement Alternat Med. 2015;2015:508958. doi: 10.1155/2015/508958. Epub 2015 Dec 22. PMID 26798398
- [Background] Kemper KJ, Heyer G, Pakalnis A, Binkley PF. What Factors Contribute to Headache-Related Disability in Teens? Pediatr Neurol. 2016 Mar;56:48-54. doi: 10.1016/j.pediatrneurol.2015.10.024. Epub 2015 Dec 24. PMID 26810775
- [Background] Leonardi M, Raggi A. A narrative review on the burden of migraine: when the burden is the impact on people's life. J Headache Pain. 2019 Apr 25;20(1):41. doi: 10.1186/s10194-019-0993-0. PMID 31023226